CLINICAL TRIAL: NCT05221814
Title: Pathological Classification of Pulmonary Nodules From Gross Images of Tumor Using Deep Learning
Brief Title: Pathological Classification of Pulmonary Nodules in Images Using Deep Learning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Collaborators: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Haiyu Zhou, vice-president, Jiangxi Provincial Cancer Hospital
Other Study IDs: 2021ky228
Record Dates: First submitted 2022-01-05; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Lung Cancer; Artificial Intelligence
Keywords: lung cancer; pathologic prediction; deep learning
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: gross pathologic photo based deep learning model — Whether apply gross pathologic photo based deep learning model to predict pathologic subtype

SUMMARY:
This study aimed to develop a deep-learning model to automatically classify pulmonary nodules based on white-light images and to evaluate the model performance. Besides, suitable operation could be chosen with the help of this model, which could shorten the time of surgery.

DETAILED DESCRIPTION:
All white-light photographs of pulmonary nodules from phones of pathologically confirmed adenocarcinoma in situ (AIS), minimally invasive adenocarcinoma (MIA) and invasive adenocarcinoma (IAC) were retrospectively collected from consecutive patients who underwent surgery between June 30, 2020 and September 15, 2021 at Guangdong Provincial People's Hospital.Finally, a total of 1037 white-light images from 973 individuals were included in the study. The entire dataset was divided into training and test datasets, which were mutually exclusive, using random sampling. Of these, 830 images were used as the training dataset and 104 images from were used as the test dataset. The CNN model was used in classifying images, namely, Resnet-50. For the CNN model, pretrained model with the ImageNet Dataset were adopted using transfer learning. After constructing the CNN models using the training dataset, the performance of the models was evaluated using the test dataset and the prospective validation dataset.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female，18 years and older.
2. Patients haven't undergone any therapy.
3. The pulmonary nodules were confirmed AIS, MIA or IAC.
4. The sizes of pulmonary nodules were less than 3cm.
5. The images were jpg format.

Exclusion Criteria:

1. Suffering from other tumor disease before or at the same time.
2. Images with poor quality or low resolution that precluded proper classification.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in Guangdong Provincial People's hospital from June 30, 2020 to September 15, 2021.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
1. Pathological subtype | through study completion, an average of 2 year
  According to WHO classification of pulmonary tumors in 2020, this study classify pulmonary tumors into adenocarcinoma in situ (AIS), minimally invasive adenocarcinoma (MIA) and invasive adenocarcinoma (IAC). We would collect the reports of pathological type of pulmonary nodules after surgery.
Area Under the Curve (AUC) | through study completion, an average of 2 year
  The area under the ROC curve based the predicton efficency of model

CONTACTS AND LOCATIONS:
Overall Officials: Haiyu Zhou, Principal Investigator — Guangdong Provincial People's Hospital
Locations (2):
- China (2):
  - Guagndong Provincial People's Hospital, Guangzhou, Guangdong
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi